CLINICAL TRIAL: NCT03260803
Title: Valuating the Effects of Oligopin Supplementation on the Turnover of Bone Formation and Antioxidant Changes in Postmenopausal Osteopenic Women: A Randomized Double-blind Clinical Trial With Placebo-concurrent Controls
Brief Title: Oligopin Supplementation and Bone Turnover Markers and Antioxidant Changes in Postmenopausal Osteopenic Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Solaleh EmamGholi, Principal Investigator, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 34606
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Osteopenia
Keywords: osteopenia; oligopin; postmenopause; antioxidant; bone
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postmenopausal osteopenic women receiveing Oligopin (Experimental): postmenopausal osteopenic women receiving Oligopin ,150 mg ,once daily, 12 week
  Interventions: Drug: Oligopin
- postmenopausal osteopenic women receiving placebo (Placebo Comparator): postmenopausal osteopenic women receiving placebo, 150 mg,once daily,12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oligopin — Oligopin ,150 mg ,once daily, 12 week
  Arms: postmenopausal osteopenic women receiveing Oligopin
Drug: Placebo — Placebo,150 mg ,once daily, 12 week
  Arms: postmenopausal osteopenic women receiving placebo

SUMMARY:
Osteoporosis fractures impose a significant economic burden on the health system. There is evidence that osteoporosis has a high prevalence in Iran (4.8% for men and 7.7% for women), and the frequency of osteopenia is 36.8% for men and 39.3% for women in Iran Accordingly, the prevention of osteopenia progression towards osteoporosis has been considered as an important issue in medicine. Bone is a dynamic tissue that is constantly being remodeled thus the equilibrium between bone formation and resorption done by simultaneously regulating osteoclasts and osteoblasts is important. Imbalance between bone deposition and resorption contributes to reducing bone mineral density and hence increasing the risk of osteoporosis

Recently, new therapies have been focused on use of medicinal herbs, especially phytochemicals. Among phytochemicals, phytonutrients, and especially polyphenols, can act both on osteoblast and on osteoclast.

Pine bark extract (oligopin) is a rich source of polyphenols that exerts strong antioxidant and anti-inflammatory activities. It has also beneficial effects on bone turnover based on in vitro studies and animal models. Investigators aimed to investigate the effects of oligopin on bone turnover markers and plasma and peripheral mononuclear cells oxidative stress in postmenopausal women with osteopenia in a double-blind randomized clinical trial. Participants are forty four women with osteopenia divided into two groups randomly (22, having oligopin, 150 mg, once daily, for 12 weeks). The 2nd group (22 women with osteopenia) receives the same amount of the placebo. At the first and the end of the study, blood sample are taken to measure in order to peripheral blood mononuclear cells isolation and plasma separation. The levels of bone alkaline phosphatase and carboxy terminal collagen type I in plasma oxidative stress markers such as total anti-oxidant capacity, malondialdehyde, and protein carbonyl were evaluated. Furthermore, oxidative stress will be evaluated in peripheral blood mononuclear cells by measurement of expression and activity of magnesium superoxide dismutase,catalase and Nuclear factor (erythroid-derived 2)-like 2.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Postmenopausal women; Aged between 50-65; Diagnosis of osteopenia based on Tscore ( -2.5 SD ≤ Tscore ≤ -1 SD); To have equal physical, pediatric and complementary therapies for at least three months before entrance to study ;Absence of history of Bone Diseases; Absence of the history of chronic diseases including cancer, diabetes, kidney failure, liver disease, systemic inflammatory diseases, degenerative joint diseases and rheumatologic disorders, primary thalassemia, hyperparathyroidism, hyperthyroidism-Cushing's, Hypercalcaemia syndrome, Hyperglycemia ;Absence of gastrointestinal disease including Crohn's disease, ulcerative colitis, celiac disease, and chronic diarrhea and gastric or duodenal ulcers treated or with a history of gastrointestinal bleeding (according to the patient's history); Absence of history of the use of drugs that affect bone metabolism and have been regularly used for at least 6 months in the past two years: such as osteoporosis drugs (bisphosphonates, estrogen receptor selective agonists / selective antagonists, alternative HRTs, PTH), diuretics, thiazides, anticonvulsants (phenytoin, phenobarbital, sodium valproate), glucocorticoids, nonsteroidal anti-inflammatory drugs such as analgesics (nonsteroidal anti-inflammatory drugs such as naproxen, aspirin and ibuprofen), cigarettes; Absence of motor disabilities, skeletal disorders, untreated psychiatric illnesses such as psychosis, Alzheimer's disease, Parkinson's disease; To accept randomization; Absence of morbid Obesity: BMI is above 40

Exclusion Criteria:

Fracture report during the study period; Unwillingness of participants to continue the project; The occurrence of any visible side effects of supplemental effects

-

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma Osteocalcin Concentration | up to third month after intervention
  Osteocalcin levels in plasma
Plasma Carboxyl terminal collagen type I Concentration | up to third month after intervention
  Carboxyl terminal collagen type I in plasma
Osteocalcin/Carboxyl terminal collagen type I ratio | up to third month after intervention
  Osteocalcin/Carboxyl terminal collagen type I ratio

SECONDARY OUTCOMES:
MnSOD activity in peripheral blood mononuclear cells | Baseline and third month after intervention
  MnSOD activity in peripheral blood mononuclear cells
Catalase activity in peripheral blood mononuclear cells | Baseline and third month after intervention
  Catalase activity in peripheral blood mono nuclear cells
MnSOD mRNA expression peripheral blood mononuclear cells | Baseline and third month after intervention
  MnSOD mRNA expression peripheral blood mononuclear cells
Catalase mRNA expression peripheral blood mononuclear cells | Baseline and third month after intervention
  Catalase mRNA expression peripheral blood mononuclear cells
NrF2 mRNA expression peripheral blood mononuclear cells | Baseline and third month after intervention
  NrF2 mRNA expression peripheral blood mononuclear cells
Plasma Malondialdehide Concentration | Baseline and third month after intervention
  Malondialdehide levels in plasma
total antioxidant capacity | Baseline and third month after intervention
  total antioxidant capacity in plasma
protein carbonyl content | Baseline and third month after intervention
  protein carbonyl content in plasma
Plasma Total thiol concentration | Baseline and third month after intervention
  Total thiol level in plasma
Catalase activity in Plasma | Baseline and third month after intervention
  Catalase activity in plasma
MnSOD activity in Plasma | Baseline and third month after intervention
  MnSOD activity in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran